CLINICAL TRIAL: NCT00600171
Title: A Randomised, Double-blind, Placebo Controlled, Parallel Group, Dose Ranging Study Evaluating the Efficacy and Safety of GW642444M Administered Once Daily Compared With Placebo for 28 Days in Adolescent and Adult Subjects With Persistent Asthma
Brief Title: Efficacy And Safety Of GW642444M Comparing Placebo In Adolescent And Adult Subjects With Persistent Asthma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2C109575
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Results first posted 2013-08-12 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: dose ranging; placebo; asthma; safety; efficacy; pharmacokinetics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo Multi dose dry powder inhlaer
  Interventions: Drug: Placebo
- GW642444M (Experimental): GW642444M
  Interventions: Drug: GW642444M

INTERVENTIONS:
Drug: GW642444M — GW642444M
  Arms: GW642444M
Drug: Placebo — Placebo mulit-dose dry powder inhaler
  Arms: Placebo

SUMMARY:
This study is designed to determine if the investigational drug is effective and safe in individuals with asthma

ELIGIBILITY:
Inclusion criteria:

* Aged 12 years of age or older at Visit 1 For sites in the following countries, subjects recruited will be ³ 18 years of age: Germany, Hungary and the Russian Federation and any other countries where local regulations or the regulatory status of study medication permit enrolment of adults only.
* Male or eligible female subjects

A female is eligible to enter and participate in the study if she is of:

Non-child bearing potential (i.e. physiologically incapable of becoming pregnant), including any female who is post-menopausal.

Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly (i.e. in accordance with the approved product label and the instructions of the physician for the duration of the study - screening to follow-up contact):

* Complete abstinence from intercourse from screening until 2 weeks after the follow-up contact; or
* Sterilisation of male partner (vasectomy with documentation of azoospermia) prior to female subject entry into the study, and this male partner is the sole partner for that subject; or
* Implants of levonorgestral inserted for at least 1 month prior to the study medication administration but not beyond the third successive year following insertion; or
* Injectable progestogen administered for at least 1 month prior to study medication administration and administered for 1 month following study completion; or
* Oral contraceptive (combined or progestogen only) administered for at least one monthly cycle prior to study medication administration; or
* Double barrier method: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository) N.B. For German sites female subjects must use a method of birth control other than the double barrier method
* An intrauterine device (IUD), inserted by a qualified physician, with published data showing that the highest expected failure rate is less than 1% per year; or
* Estrogenic vaginal ring inserted for at least 1 month prior to study medication administration; or
* Percutaneous contraceptive patches in place for at least 1 month prior to study medication administration Female subjects should not be enrolled if they are pregnant, or lactating, or plan to become pregnant during the time of study participation.
* Documented clinical history of persistent asthma, as defined by the National Institutes of Health [NIH, 2007] first diagnosed at least 6 months prior to Visit 1.
* Subjects with current reversible airways disease as demonstrated at Visit 1 by an increase in FEV1 of ≥ 12% and ≥ 200ml over the pre-salbutamol/albuterol FEV1 at approximately 30 minutes after the inhalation of 400mcg of salbutamol/albuterol via MDI (spacer permitted for reversibility testing only if required) or one nebulised salbutamol/albuterol solution.
* Subjects must be using an inhaled corticosteroid and have been maintained on a stable dose for 4 weeks prior to Visit 1 at one of the following doses:

Maximum Allowable Concurrent Inhaled Corticosteroid Doses

Asthma Therapy(Maximum Daily Dose (mcg/day)) fluticasone propionate MDI CFC/HFA (≤ 880mcg1/ ≤1000mcg2) fluticasone propionate DPI(≤ 1000mcg) beclomethasone dipropionate(≤ 1680mcg1/ ≤ 2000mcg2) beclomethasone dipropionate HFA (QVAR)(≤ 640mcg1/ ≤ 800mcg2) budesonide DPI/MDI(≤ 2000mcg) Flunisolide(≤ 2000mcg) triamcinolone acetonide(≤ 2000mcg) mometasone furoate(≤ 880mcg) Ciclesonide(≤ 320mcg1/ ≤ 400mcg2)

CFC=chlorofluorocarbon HFA=hydrofluoroalkane

1. Ex-actuator dose
2. Ex-valve dose

   * Pre-bronchodilator FEV1 between ≥ 40 - ≤ 90% predicted at Visit 1. NHANES III predicted values will be used for subjects aged ≥ 12 years and adjustments to predicted values will be made for African American subjects [Hankinson, 1999].
   * Appropriately signed and dated informed consent has been obtained.
   * Capable of withholding salbutamol/albuterol use for ≥ 6 hours prior to clinic visits.
   * In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion criteria:

* An exacerbation of asthma within 4 weeks of Visit 1, or a culture documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear within 4 weeks of Visit 1 that led to a change in asthma management, or in the opinion of the Investigator is expected to affect the subjects asthma status or the subjects ability to participate in the study.
* History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnoea, respiratory arrest or hypoxia seizures.
* Asthma exacerbation requiring treatment with oral corticosteroids within 3 months prior to Visit 1.
* Hospitalised for an asthma exacerbation within 6 months of Visit 1. Hospitalisation is defined as an overnight stay in a hospital.
* Previously enrolled in this study, or has participated in any study using an investigational drug during the previous 30 days or will participate simultaneously in another clinical trial.
* A subject must not have any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the subject's safety at risk through study participation or would confound the interpretation of the efficacy results if the condition/disease exacerbated during the study.

The list of additional excluded conditions/diseases includes, but is not limited to the following:

congestive heart failure, known aortic aneurysm clinically significant coronary heart disease, clinically significant cardiac arrhythmia stroke within 3 months of Visit 1, uncontrolled hypertension1 poorly controlled peptic ulcer, haematologic, hepatic, or renal disease immunologic compromise, current malignancy2 tuberculosis (current or untreated3), Cushing's disease Addison's disease, uncontrolled diabetes mellitus uncontrolled thyroid disorder, recent history of drug or alcohol abuse neurological disease, pulmonary disease4

1. systolic blood pressure 160, or diastolic blood pressure >100
2. history of malignancy is acceptable only if subject has been in remission for one year prior to Visit 1 (remission = no current evidence of malignancy and no treatment for the malignancy in the 12 months prior to Visit 1)
3. Subjects with a history of tuberculosis who have received an approved prophylactic treatment regimen or an approved active treatment regimen and who have no evidence of active disease for a minimum of 2 years may be enrolled [American Thoracic Society Documents, 2005] [American Thoracic Society (ATS), 2003]
4. Including but not limited to chronic bronchitis, emphysema, bronchiectasis with the need of treatment, cystic fibrosis, bronchopulmonary dysplasia, and chronic obstructive pulmonary disease.

   * Any adverse reaction including immediate or delayed hypersensitivity to any ß2-agonist or sympathomimetic drug, or known (i.e., patients with a history of severe milk protein allergy) or suspected sensitivity to the constituents of GW642444M inhalation powder (e.g., lactose or magnesium stearate).
   * Subjects who are likely to be non-compliant with study medication and other study-related requirements (e.g. attendance at clinic visits or completion of Daily Diary).
   * Neurological or psychiatric disease or history of drug or alcohol abuse which would interfere with the subject's proper completion of the protocol requirements.

Abuse of alcohol is defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males) or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). The number of units of alcohol in a drink can be determined by multiplying the volume of the drink (in millilitres) by its percentage ABV and dividing by 1000

* Current smoker or a smoking history of 10 pack years or more (e.g. 20 cigarettes/day for 10 years). A subject may not have used tobacco products within the past one year (i.e., cigarettes, cigars, or pipe tobacco).
* Administration of systemic, oral or depot corticosteroids or administration of anti-IgE (e.g. omalizumab [Xolair]) within 12 weeks of Visit 1.
* Administration of the following asthma medications within 14 days of Visit 1:
* Theophyllines
* Oral β2-agonists (e.g. bambuterol)
* Slow-release bronchodilators
* Anticholinergics - short or long-acting
* Oral long acting antihistamines
* Oral leukotriene receptor antagonists (e.g. montelukast)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (81):
- United States (28):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Valrico, Florida
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, River Forest, Illinois
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Skillman, New Jersey
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
- Argentina (4):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Mendoza, Mendoza Province
  - GSK Investigational Site, San Miguel de Tucumán
- Belgium (2):
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Liège
- Canada (6):
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Chile (2):
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- France (3):
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
- Germany (8):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Wiesloch, Baden-Wurttemberg
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- Netherlands (3):
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Utrecht
- Peru (2):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Lima
- Philippines (2):
  - GSK Investigational Site, Cavite
  - GSK Investigational Site, Manila
- Poland (4):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
- Russia (6):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Yaroslavl
- South Africa (5):
  - GSK Investigational Site, Cape Town, Gauteng
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Claremont
  - GSK Investigational Site, eManzimtoti
  - GSK Investigational Site, Mowbray
- South Korea (2):
  - GSK Investigational Site, Cheongju, Chungcheongbuk-do
  - GSK Investigational Site, Suwon
- Sweden (2):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Lund
- Thailand (2):
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Lotvall J, Bateman ED, Bleecker ER, Busse WW, Woodcock A, Follows R, Lim J, Stone S, Jacques L, Haumann B. 24-h duration of the novel LABA vilanterol trifenatate in asthma patients treated with inhaled corticosteroids. Eur Respir J. 2012 Sep;40(3):570-9. doi: 10.1183/09031936.00121411. Epub 2012 Feb 23. PMID 22362859
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: B2C109575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: B2C109575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: B2C109575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: B2C109575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: B2C109575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: B2C109575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: B2C109575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 614 participants were randomized to study drug; however, 7 of these participants were randomized in error and did not receive any study drug. 607 participants comprised the Intent-to-Treat Population (all participants randomized to treatment and who received at least one dose of study medication).
Pre-assignment Details: Participants were screened (Visit 1), for eligibility, which included the inhaled albuterol/salbutamol reversibility test. Following screening and a 14-day Run-in period, participants meeting eligibility criteria were stratified in an approximately 1:1 ratio according to their Baseline Forced Expiratory Volume per one second (FEV1).
Groups:
- Placebo: Particpants received placebo at the clinic on Days 1 7, 14, and 28, and self-administered placebo on non-clinic study days, once daily in the evening via the Dry Powder Inhaler (DPI). Participants remained on their current ICS therapy (at fixed doses) throughout the study (screening to follow-up inclusive).
- GW642444M 3 µg: Particpants received GW642444M 3 micrograms (µg) at the clinic on Days 1, 7, 14, and 28, and self administered GW642444M 3 µg on non-clinic study days, once daily in the evening via the DPI. Participants remained on their current ICS therapy (at fixed doses) throughout the study (screening to follow-up inclusive).
- GW642444M 6.25 µg: Particpants received GW642444M 6.25 µg at the clinic on Days 1, 7, 14, and 28, and self administered GW642444M 6.25 µg on non-clinic study days, once daily in the evening via the DPI. Participants remained on their current ICS therapy (at fixed doses) throughout the study (screening to follow-up inclusive).
- GW642444M 12.5 µg: Particpants received GW642444M 12.5 µg at the clinic on Days 1, 7, 14, and 28, and self administered GW642444M 12.5 µg on non-clinic study days, once daily in the evening via the DPI. Participants remained on their current ICS therapy (at fixed doses) throughout the study (screening to follow-up inclusive).
- GW642444M 25 µg: Particpants received GW642444M 25 µg at the clinic on Days 1, 7, 14, and 28, and self administered GW642444M 25 µg on non-clinic study days, once daily in the evening via the DPI. Participants remained on their current ICS therapy (at fixed doses) throughout the study (screening to follow-up inclusive).
- GW642444M 50 µg: Particpants received GW642444M 50 µg at the clinic on Days 1, 7, 14, and 28, and self administered GW642444M 50 µg on non-clinic study days, once daily in the evening via the DPI. Participants remained on their current ICS therapy (at fixed doses) throughout the study (screening to follow-up inclusive).
Period: Overall Study
Arm/Group | Placebo | GW642444M 3 µg | GW642444M 6.25 µg | GW642444M 12.5 µg | GW642444M 25 µg | GW642444M 50 µg
Started | 102 | 101 | 101 | 100 | 101 | 102
Completed | 86 | 84 | 91 | 88 | 93 | 97
Not Completed | 16 | 17 | 10 | 12 | 8 | 5
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 9 | 12 | 3 | 5 | 4 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 1 | 0 | 0
Not completed — Met Protocol-defined Stopping Criteria | 3 | 1 | 7 | 3 | 2 | 2
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GW642444M 3 µg | GW642444M 6.25 µg | GW642444M 12.5 µg | GW642444M 25 µg | GW642444M 50 µg | Total
Number analyzed (Participants) | 102 | 101 | 101 | 100 | 101 | 102 | 607
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.9 (15.60) | 44.4 (13.50) | 42.4 (14.13) | 41.3 (15.33) | 42.2 (14.27) | 44.0 (15.22) | 42.4 (14.72)
Gender [Count of Participants; unit: Participants]
  Female | 61 | 52 | 51 | 56 | 61 | 57 | 338
  Male | 41 | 49 | 50 | 44 | 40 | 45 | 269
Race/Ethnicity, Customized [Number; unit: participants]
  African American (AfAm)/African Heritage (AfH) | 4 | 11 | 8 | 12 | 14 | 8 | 57
  American Indian (AmIn) or Alaska Native (AN) | 3 | 2 | 3 | 2 | 2 | 1 | 13
  Central/South Asian Heritage (Her) | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Japanese/East Asian (EA) Her/South EA Her | 10 | 13 | 11 | 8 | 8 | 9 | 59
  Native Hawaiian or other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 81 | 74 | 77 | 75 | 75 | 83 | 465
  AfAm/AfH & AmIn or AN | 0 | 1 | 0 | 0 | 0 | 0 | 1
  AfAm/AfH & White | 2 | 0 | 0 | 0 | 0 | 0 | 2
  AmIn or AN & White | 1 | 0 | 1 | 2 | 1 | 1 | 6
  Asian & White | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Clinic Visit Trough FEV1 at Day 28 (Last Observation Carried Forward [LOCF])
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1), defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 is defined as the clinic visit (pre-bronchodilator and pre-dose) FEV1 at the end of the 28-day treatment period, with the trough FEV1 defined as the mean of the 23 hour and 24 hour post-dose assessments on Day 28. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Analysis was performed using Analysis of Covariance (ANCOVA) using LOCF with covariates of Baseline (pre-dose on Day 1), country, sex, age, stratum, and treatment.
Time Frame: Baseline and Day 28
Population: ITT Population: all participants who were randomized to treatment and received at least one dose of study medication. The LOCF method was used to impute missing data. When the endpoint was missing, the last valid non-missing on-treatment, post-Baseline trough assessment was used instead. Only measurements from scheduled visits were used.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | GW642444M 3 µg | GW642444M 6.25 µg | GW642444M 12.5 µg | GW642444M 25 µg | GW642444M 50 µg
Number analyzed (Participants) | 95 | 98 | 99 | 97 | 99 | 100
Liters | 0.147 (0.036) | 0.212 (0.036) | 0.217 (0.035) | 0.278 (0.036) | 0.269 (0.035) | 0.309 (0.035)
Statistical Analysis 1: Comparison: Placebo vs GW642444M 3 µg; Test type: Superiority or Other; p = 0.208, ANCOVA; Mean Difference (Final Values) = 0.064, 95% CI 2-sided [-0.036 to 0.164]
Statistical Analysis 2: Comparison: Placebo vs GW642444M 6.25 µg; Test type: Superiority or Other; p = 0.169, ANCOVA; Mean Difference (Final Values) = 0.069, 95% CI 2-sided [-0.029 to 0.168]
Statistical Analysis 3: Comparison: Placebo vs GW642444M 12.5 µg; Test type: Superiority or Other; p = 0.011, ANCOVA; Mean Difference (Final Values) = 0.130, 95% CI 2-sided [0.030 to 0.230]
Statistical Analysis 4: Comparison: Placebo vs GW642444M 25 µg; Test type: Superiority or Other; p = 0.016, ANCOVA; Median Difference (Final Values) = 0.121, 95% CI 2-sided [0.023 to 0.220]
Statistical Analysis 5: Comparison: Placebo vs GW642444M 50 µg; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = 0.162, 95% CI 2-sided [0.062 to 0.261]

2. Secondary Outcome: Mean Change From Baseline in Clinic Visit Trough FEV1 at Day 28 Per Stratum (LOCF)
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1), defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 is defined as the clinic visit (pre-bronchodilator and pre-dose) FEV1 at the end of the 28-day treatment period, with the trough FEV1 defined as the mean of the 23 hour and 24 hour post-dose assessments on Day 28. Change from Baseline in trough FEV1 at the end of the treatment period (23 hours and 24 hours after dosing on Day 28) was analyzed for each stratum (Lower stratum: FEV1 percent predicted, >=40% to <=65%; Upper stratum: FEV1 percent predicted, >=65% to <=90%). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Analysis was performed using ANCOVA using LOCF with covariates of Baseline (pre-dose on Day 1), country, sex, age, stratum, treatment, and treatment by stratum interaction.
Time Frame: Baseline and Day 28
Population: ITT Population. The LOCF method was used to impute missing data. When the endpoint was missing, the last valid non-missing on-treatment, post-Baseline trough assessment was used instead. Only measurements from scheduled visits were used. Only those participants with available data (using LOCF) at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- GW642444M 12.5 µg: Particpants received GW642444M 12.5 µg at the clinic on Days 1, 7, 14, and 28, and self administered GW642444M 12.5 µgon non-clinic study days, once daily in the evening via the DPI. Participants remained on their current ICS therapy (at fixed doses) throughout the study (screening to follow-up inclusive).
Arm/Group | Placebo | GW642444M 3 µg | GW642444M 6.25 µg | GW642444M 12.5 µg | GW642444M 25 µg | GW642444M 50 µg
Number analyzed (Participants) | 95 | 98 | 99 | 97 | 99 | 100
Liters
  Lower stratum, n=43, 44, 41, 40, 46, 45 | 0.210 (0.057) | 0.161 (0.056) | 0.247 (0.057) | 0.319 (0.057) | 0.281 (0.054) | 0.349 (0.055)
  Upper stratum, n=52, 54, 58, 57, 53, 55 | 0.098 (0.049) | 0.254 (0.051) | 0.194 (0.048) | 0.247 (0.049) | 0.259 (0.049) | 0.276 (0.049)

3. Secondary Outcome: Change From Baseline in Weighted Mean 24-hour Serial FEV1 at Day 1 and Day 28
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Change from Baseline in weighted mean for 24-hour serial FEV1 on Days 1 and Day 28 was assessed. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline (pre-dose on Day 1), country, sex, age, stratum, and treatment.
Time Frame: Baseline; Day 1 and Day 28 (mean post-dose FEV1 after 15, 30, and 60 minutes and 2, 3, 4, 6, 12, 16, 20, 22, 23, and 24 hours)
Population: ITT Population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | GW642444M 3 µg | GW642444M 6.25 µg | GW642444M 12.5 µg | GW642444M 25 µg | GW642444M 50 µg
Number analyzed (Participants) | 101 | 100 | 101 | 99 | 100 | 100
Liters
  Day 1, n=101, 100, 101, 99, 100, 100 | 0.137 (0.029) | 0.239 (0.029) | 0.215 (0.029) | 0.267 (0.029) | 0.330 (0.029) | 0.352 (0.029)
  Day 28, n=87, 83, 91, 88, 93, 97 | 0.149 (0.032) | 0.300 (0.033) | 0.253 (0.031) | 0.292 (0.032) | 0.315 (0.031) | 0.321 (0.031)

4. Secondary Outcome: Mean Change From Baseline in Trough (Pre-dose and Pre-bronchodilator) Daily Evening (PM) Peak Expiratory Flow (PEF) Averaged Over the 28-day Treatment Period
Description: Peak Expiratory Flow (PEF) is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. Change from Baseline was calculated as the value of the averaged PEF daily PM over the 28-day treatment period (at Day 28) minus the Baseline value (defined as the last 7 days prior to randomization of the participants). Analysis was performed using ANCOVA with covariates of Baseline, country, sex, age, stratum, and treatment.
Time Frame: Baseline and Days 1-28
Population: ITT Population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | Placebo | GW642444M 3 µg | GW642444M 6.25 µg | GW642444M 12.5 µg | GW642444M 25 µg | GW642444M 50 µg
Number analyzed (Participants) | 99 | 99 | 101 | 98 | 101 | 102
Liters per minute | 0.4 (3.87) | 14.0 (3.87) | 24.5 (3.82) | 28.9 (3.87) | 34.0 (3.81) | 38.4 (3.82)

5. Secondary Outcome: Mean Change From Baseline in Daily Morning (AM) PEF Averaged Over the 28-day Treatment Period
Description: Peak Expiratory Flow (PEF) is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. Change from Baseline was calculated as the value of the averaged PEF daily AM over the 28-day treatment period (at Day 28) minus the Baseline value (defined as the last 7 days prior to randomization of the participants). Analysis was performed using ANCOVA with covariates of Baseline, country, sex, age, stratum, and treatment.
Time Frame: Baseline and Days 1-28
Population: ITT Population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Groups:
- GW642444M 6.25 µg: Particpants received GW642444M 6.25 µg at the clinic on Days 1, 7, 14, and 28, and self administered GW642444M 6.25 µg µgon non-clinic study days, once daily in the evening via the DPI. Participants remained on their current ICS therapy (at fixed doses) throughout the study (screening to follow-up inclusive).
Arm/Group | Placebo | GW642444M 3 µg | GW642444M 6.25 µg | GW642444M 12.5 µg | GW642444M 25 µg | GW642444M 50 µg
Number analyzed (Participants) | 98 | 99 | 101 | 98 | 101 | 102
Liters per minute | 1.9 (3.69) | 18.7 (3.67) | 26.8 (3.63) | 34.2 (3.68) | 38.1 (3.61) | 44.0 (3.63)

6. Secondary Outcome: Mean Change From Baseline in the Percentage of Symptom-free 24-hour (hr) Periods Averaged Over the 28-day Treatment Period
Description: Participants who were symptom free for 24 hours were assessed. Change from Baseline was calculated as the value at Day 28 minus the value at Baseline (defined as the last 7 days prior to randomization of the participants). Analysis was performed using ANCOVA with covariates of Baseline, country, sex, age, stratum, and treatment.
Time Frame: Baseline and Days 1-28
Population: ITT Population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free 24-hr periods
Arm/Group | Placebo | GW642444M 3 µg | GW642444M 6.25 µg | GW642444M 12.5 µg | GW642444M 25 µg | GW642444M 50 µg
Number analyzed (Participants) | 98 | 99 | 101 | 98 | 101 | 102
Percentage of symptom-free 24-hr periods | 14.2 (3.27) | 22.6 (3.25) | 23.6 (3.21) | 26.8 (3.26) | 36.4 (3.21) | 32.3 (3.21)

7. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free 24-hour (hr) Periods Averaged Over the 28-day Treatment Period
Description: The time span during which the participants did not have to take any rescue medication (medication intended to relieve symptoms immediately) was considered to be a rescue-free period. Change from Baseline is calculated as the value at Day 28 minus the value at Baseline (defined as the last 7 days prior to randomization of the participants). Analysis was performed using ANCOVA with covariates of Baseline, country, sex, age, stratum, and treatment.
Time Frame: Baseline and Days 1-28
Population: ITT Population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free 24-hr periods
Arm/Group | Placebo | GW642444M 3 µg | GW642444M 6.25 µg | GW642444M 12.5 µg | GW642444M 25 µg | GW642444M 50 µg
Number analyzed (Participants) | 99 | 99 | 101 | 98 | 101 | 102
Percentage of rescue-free 24-hr periods | 15.0 (3.33) | 25.8 (3.33) | 27.3 (3.28) | 29.6 (3.34) | 43.4 (3.28) | 34.0 (3.28)

8. Secondary Outcome: Difference in Post Salbutamol/Albuterol FEV1 (FEV1 30 Minutes After a Single Dose of 400 µg Salbutamol/Albuterol) Between the Following Time Points: 24 Hours After Dosing on Day 1 and Day 28
Description: Assessment at Visit 2/2a was made prior to the evening dose of study medication on Day 2. Participants were administered a single 400 µg dose of salbutamol/albuterol, and FEV1 was measured 30 minutes after this administration. The highest of three technically acceptable measurements was recorded. These assessments were performed as follows: between 5 PM and 10 PM, >=6 hours after the last use of salbutamol/albuterol, >=6 hours after the last caffeine consumption, >=2 hours after exercise (or strenuous activity), >=24 hours after the first dose (Visit 2) or last dose (Visit 5) of study medication. Analysis was performed using ANCOVA with covariates of Baseline (pre-salbutamol measurement at Screening), country, sex, age, stratum, and treatment. Analysis is of the differences in absolute FEV1 measurements taken post-salbutamol/albuterol.
Time Frame: 24 hours after dosing on Day 1 (Visit 2) and on Day 28 (Visit 5)
Population: ITT Population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | GW642444M 3 µg | GW642444M 6.25 µg | GW642444M 12.5 µg | GW642444M 25 µg | GW642444M 50 µg
Number analyzed (Participants) | 83 | 80 | 87 | 86 | 86 | 92
Liters | -0.039 (0.023) | -0.035 (0.024) | -0.012 (0.023) | -0.017 (0.023) | -0.062 (0.023) | -0.049 (0.022)

9. Secondary Outcome: Difference in Post Salbutamol/Albuterol FEV1 (FEV1 30minutes After a Single Dose of 400 µg Salbutamol/Albuterol) Between the Following Time Points: Screening and 24 Hours After Dosing on Day 1
Description: Assessment at Visit 2/2a was made prior to the evening dose of study medication on Day 2. Participants were administered a single 400 µg dose of salbutamol/albuterol, and FEV1 was measured 30 minutes after this administration. The highest of three technically acceptable measurements was recorded. These assessments were performed as follows: between 5 PM and 10 PM, >=6 hours after the last use of salbutamol/albuterol, >=6 hours after the last caffeine consumption, >=2 hours after exercise (or strenuous activity), Screening and >=24 hours after the first dose (Visit 2) of study medication. Analysis was performed using ANCOVA with covariates of Baseline (pre-salbutamol measurement at Screening), country, sex, age, stratum, and treatment. Analysis is of the differences in absolute FEV1 measurements taken post-salbutamol/albuterol.
Time Frame: Screening (Visit 1) and 24 hours after dosing on Day 1 (Visit 2)
Population: ITT Population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | GW642444M 3 µg | GW642444M 6.25 µg | GW642444M 12.5 µg | GW642444M 25 µg | GW642444M 50 µg
Number analyzed (Participants) | 97 | 97 | 98 | 99 | 96 | 98
Liters | -0.040 (0.028) | 0.008 (0.028) | -0.061 (0.028) | -0.029 (0.028) | -0.020 (0.028) | -0.060 (0.028)

10. Secondary Outcome: Difference in Post Salbutamol/Albuterol FEV1 (FEV1 30 Minutes After a Single Dose of 400 µg Salbutamol/Albuterol) Between the Following Time Points: Screening and 24 Hours After Dosing on Day 28
Description: as for outcome 9
Time Frame: Screening (Visit 1) and 24 hours after dosing on Day 28 (Visit 5)
Population: ITT Population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | GW642444M 3 µg | GW642444M 6.25 µg | GW642444M 12.5 µg | GW642444M 25 µg | GW642444M 50 µg
Number analyzed (Participants) | 84 | 80 | 89 | 86 | 88 | 93
Liters | -0.076 (0.031) | -0.022 (0.031) | -0.055 (0.030) | -0.048 (0.030) | -0.086 (0.030) | -0.104 (0.029)

ADVERSE EVENTS:
Time Frame: On-treatment adverse events (AEs), defined as those events occurring while participants were on treatment, up to and including the day after the last dose in each treatment period (up to Day 28), are reported.
Description: Serious adverse events (SAEs) and non-serious AEs were collected in the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of study medication.
Arm/Group | Placebo | GW642444M 3 µg | GW642444M 6.25 µg | GW642444M 12.5 µg | GW642444M 25 µg | GW642444M 50 µg
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/101 | 0/101 | 0/100 | 0/101 | 0/102
Other Adverse Events (participants affected / at risk) | 14/102 | 15/101 | 9/101 | 12/100 | 9/101 | 11/102
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=102) | GW642444M 3 µg (N=101) | GW642444M 6.25 µg (N=101) | GW642444M 12.5 µg (N=100) | GW642444M 25 µg (N=101) | GW642444M 50 µg (N=102)
Headache (Nervous system disorders) | 8 | 12 | 7 | 9 | 7 | 8
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1 | 3 | 2 | 2
Nasopharyngitis (Infections and infestations) | 4 | 2 | 2 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.